CLINICAL TRIAL: NCT01174472
Title: Drug Eluting Versus Conventional Balloon Angioplasty for the Treatment of Failing Dialysis Access. A Prospective Randomized Single-Center Trial.
Brief Title: Drug Eluting Balloon Angioplasty for Dialysis Access Treatment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, SIABLIS DIMITRIOS, Professor of Radiology, University of Patras
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9462/14-4-2010
Record Dates: First submitted 2010-07-21; First posted 2010-08-03 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2012-01

CONDITIONS: Dialysis; Angioplasty
Keywords: Dialysis access; angioplasty; drug eluting balloon
MeSH Terms: interventions — Angioplasty

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Balloon Angioplasty (COBA) (Active Comparator): Patients with lesions treated with conventional balloon angioplasty
  Interventions: Device: Percutaneous Transluminal Angioplasty (PTA)
- Drug Eluting Balloon Angioplasty (DEB) (Experimental): Patients with lesions treated with Drug Balloon Angioplasty
  Interventions: Device: Percutaneous Transluminal Angioplasty (PTA)

INTERVENTIONS:
Device: Percutaneous Transluminal Angioplasty (PTA) — Angioplasty performed with the use of the novel paclitaxel eluting balloons
  Other Names: IN.PACT ADMIRAL, Paclitaxel eluting dilatation PTA catheter
  Arms: Drug Eluting Balloon Angioplasty (DEB)
Device: Percutaneous Transluminal Angioplasty (PTA) — Angioplasty performed with the use of conventional angioplasty balloons
  Other Names: Conquest PTA Balloon Dilatation Catheter
  Arms: Conventional Balloon Angioplasty (COBA)

SUMMARY:
The aim of the study is to compare the feasibility and the effectiveness, by means of immediate and long-term results, of drug eluting balloon (DEB) versus conventional balloon angioplasty for the treatment of failing dialysis access.

DETAILED DESCRIPTION:
In total 40 patients already diagnosed with hemodynamically significant stenosis of the dialysis AVF or AVG (including venous outflow lesions), programmed to undergo percutaneous transluminal angioplasty by our department, will sign informed consent and will be randomized to either receive DEB (Paclitaxel eluting balloon), or conventional balloon therapy. The protocol includes the description of patient's demographics (age, gender,dialysis access details, risk factors) and procedural details, as well as immediate results and long-term follow up.

ELIGIBILITY:
Inclusion Criteria:

* Angiographic and clinical diagnosis of dysfunctional dialysis access due to one or more stenotic lesions.
* Patients with AVF or AVG
* Fistula or graft or vessel diameter ranging from 3 mm up to 12 mm

Exclusion Criteria:

* Fistula or graft or vessel diameter < 3 mm and > 12 mm
* History of severe allergic reaction to contrast media
* Intolerance to aspirin and/or clopidogrel
* Systemic coagulopathy or hypercoagulation disorders

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-03; Primary Completion 2010-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Technical success | 1 minute after the final balloon angioplasty
  Residual stenosis of the treated lesion less than 30%, without any hemodynamicaly significant dissection (Type C)after the final angiography
Primary patency | 1 year
  Angiographic visualization of a lesion with <50% restenosis and no need for any additional repeat interventional procedure within the previously treated lesion, due to failing access.

SECONDARY OUTCOMES:
Secondary patency | 1 year
  Angiographicaly proven patency (<50% restenosis and no need for any additional repeat interventional procedure within the previously treated lesion, due to failing access)of the treated lesion following one re-intervention procedure of any kind.
Target lesion re-intervention (TLR)-free interval | 1 year
  The time interval without any additional recanalization procedure within the area of the treated lesion, because of angiographic or/and clinical deterioration
Major complications rates | Periprocedural and up to 1 year
  Classified according to published international guidelines and reporting standards
Minor complications rates | Periprocedural and up to 1 year follow-up
  Classified according to published international guidelines and reporting standards

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Siablis, MD, PhD, Principal Investigator — University Hospital of Patras
Locations (1):
- Patras University Hospital, Department of Radiology, Angiography Suite, Rio, Achaias, Greece

REFERENCES:
- [Derived] Kitrou PM, Katsanos K, Spiliopoulos S, Karnabatidis D, Siablis D. Drug-eluting versus plain balloon angioplasty for the treatment of failing dialysis access: final results and cost-effectiveness analysis from a prospective randomized controlled trial (NCT01174472). Eur J Radiol. 2015 Mar;84(3):418-423. doi: 10.1016/j.ejrad.2014.11.037. Epub 2014 Dec 15. PMID 25575743
- [Derived] Katsanos K, Karnabatidis D, Kitrou P, Spiliopoulos S, Christeas N, Siablis D. Paclitaxel-coated balloon angioplasty vs. plain balloon dilation for the treatment of failing dialysis access: 6-month interim results from a prospective randomized controlled trial. J Endovasc Ther. 2012 Apr;19(2):263-72. doi: 10.1583/11-3690.1. PMID 22545894